CLINICAL TRIAL: NCT00004705
Title: Study of Uridine Triphosphate (UTP) as an Aerosol Spray for Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: University of North Carolina (Other)
Purpose: Treatment
Other Study IDs: 199/13446; UNCCH-FDR001008
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Amiloride; Uridine

INTERVENTIONS:
Drug: amiloride
Drug: uridine

SUMMARY:
OBJECTIVES: I. Determine the stability of uridine triphosphate (UTP) and examine the metabolism of exogenous nucleotides on airway epithelial surfaces in patients with cystic fibrosis.

II. Determine the acute safety and efficacy of aerosolized UTP in children with cystic fibrosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients may be treated on any of three different regimens. Patients may be treated on more than one regimen, if they meet the eligibility requirements.

Patients on regimen A are adults and receive uridine triphosphate (UTP) by inhalation, followed immediately by bronchoscopy.

Patients on regimen B are children, aged 4 to 10 years. Patients receive up to 4 graded doses of UTP by inhalation on day 1. On day 2, patients receive a single dose of UTP. Patients receive amiloride followed by UTP by inhalation on day 3.

Patients on regimen C are children, aged 4 to 18 years. Patients inhale a radiolabelled (technetium 99m) monodisperse iron oxide aerosol. Radiation deposited in the patient's lungs is monitored. Patients are randomized to receive one of 4 different aerosols (vehicle; UTP; amiloride; or UTP plus amiloride), which is inhaled for 20 minutes. Patients are followed 24 hours after aerosol exposure.

Regimen D is a dose escalation study in which patients are aged 9 to 40 years. Patients receive either the vehicle or UTP by inhalation 3 times daily for 3 days. Cohorts of 4 patients each are entered at each dose level.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of mild to moderate cystic fibrosis Small production of daily airway secretions Stable pulmonary course --Prior/Concurrent Therapy-- Radiotherapy: No radiation within 12 months to cause patient to exceed annual limits Other: No chronic medication for reactive airways disease At least 12 hours since inhaled beta-adrenergic agonists At least 24 hours since systemic theophylline --Patient Characteristics-- FEV1 greater than 50% predicted Other: Not pregnant Must perform reproducible spirometry

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Knowles, Study Chair — University of North Carolina